CLINICAL TRIAL: NCT03839524
Title: A Phase I Trial Evaluating a Mutanome-directed Immunotherapy in Patients With High Grade Serous Carcinoma (HGSC) of the Ovary, Fallopian Tube or Peritoneum.
Brief Title: A Trial Evaluating TG4050 in Ovarian Carcinoma.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Transgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG4050.01
Record Dates: First submitted 2019-02-06; First posted 2019-02-15 (Actual); Results first posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Ovarian Carcinoma; Fallopian Tube Cancer; Peritoneal Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TG4050 arm (Experimental): Patients in this arm will receive injections of TG4050 Investigational Medicinal Product.
  Interventions: Drug: TG4050

INTERVENTIONS:
Drug: TG4050 — Subcutaneous injections weekly for the first 6 weeks and then every 3 weeks.

SUMMARY:
This is a multicenter, open-label, single arm phase I study evaluating the safety and tolerability as well as some activity parameters of TG4050 in patients with ovarian, fallopian or peritoneal serous carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Female patients ≥ 18 years
3. Histologically confirmed high grade, advanced stage serous ovarian, fallopian tube or primary peritoneal carcinoma.
4. Patients who have undergone primary debulking surgery or interval debulking surgery and have completed standard first-line platinum-based chemotherapy and for whom tumor tissue has been banked.
5. Patients must have achieved a complete response to therapy
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at treatment period initiation
7. Adequate hematological, hepatic and renal functions.

Exclusion Criteria:

1. Patient having received any cancer immunotherapy including cancer vaccines, any antibody/drug targeting T cell co-regulatory proteins such as anti-Programmed cell death 1 (anti-PD1), anti-Programmed death-ligand 1 (anti-PDL1) or anti-cytotoxic T-lymphocyte-associated protein 4 (anti-CTL4)
2. Patients with other active malignancy ≤ 3 years prior to registration except non-melanoma skin cancer, stage 0 in situ carcinoma.
3. Patient post-organ transplantation, including allogeneic stem cell or bone marrow transplantation.
4. Known history of positive testing for Human Immunodeficiency Virus (HIV) or known AIDS (Acquired Immune Deficiency Syndrome).
5. Any known allergy or reaction to eggs or attributed to compounds of similar chemical or biological composition to therapeutic vaccines/immunotherapeutic products.
6. Acute or chronic infection with hepatitis C Virus (HCV) or Hepatitis B Virus (HBV).
7. Major surgery within 4 weeks of treatment start.
8. Treatment with another investigation agent within 30 days prior to TG4050 treatment initiation.
9. Patients under chronic treatment with systemic corticosteroids or other immunosuppressive drugs . Steroids with no or minimal systemic effect (topical, inhalation) are allowed.
10. Use of live vaccine for the prevention of infectious diseases during the four-week period prior to TG4050 treatment initiation planned date. Furthermore, patients should not receive any live vaccine during the period of study treatment administration.
11. Uncontrolled intercurrent illness.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (3):
  - Mayo Clinic Phoenix, Phoenix, Arizona
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Mayo Clinic Rochester, Rochester, Minnesota
- France (3):
  - Institut Curie, Paris
  - Hôpital Pitié-Salpêtrière, Paris
  - IUCT Toulouse, Toulouse

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 64 patients consented to participate in the study. Of these, 58 (90.6%) were non-included-21 at study entry and 37 at baseline-while 6 patients were assigned to treatment.
Groups:
- TG4050 Arm: Participants received subcutaneous injections of TG4050 at a dose of 1 × 10⁸ PFU weekly for the first six weeks, and then every three weeks, for up to a maximum of 20 injections.
  As only one participant was treated in Cohort A (no measurable disease at treatment initiation), the results are presented by combining both cohorts, for a total of six participants.
Period: Overall Study
Arm/Group | TG4050 Arm
Started | 6
Completed | 5
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | TG4050 Arm
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 5
Age, Continuous [Median (Full Range); unit: years] | 73.5 [47 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 5
  France | 1
BMI [Mean (Standard Deviation); unit: kg/m²] | 29.3 (4.79)
Eastern Cooperative Oncology Group Performance Status (ECOG PS) [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) score is an overall assessment of the functional/physical performance of the patient.
  0=Fully active, able to carry on all pre-disease performance without restriction. 1=Restricted in strenuous activity but ambulatory and able to carry out work of a sedentary nature.
  Participants
    ECOG status 0 | 5
    ECOG status 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability (Adverse Event Reported Per CTCAE v5)
Description: Incidence of Adverse Events as assessed by the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0
Time Frame: Up to 1 year . Adverse events were collected from treatment initiation weekly for the first six weeks, every three weeks thereafter until 30 days after the last treatment administration.
Population: Safety Analysis Set (SAF): all patients included and who received at least one dose of TG4050.
Measure: Count of Participants; unit: Participants
Arm/Group | TG4050 Arm
Number analyzed (Participants) | 6
Participants
  Adverse Event | 6
  Dose Limiting Toxicity | 0
  AE related to TG4050 | 6
  Injection site reaction | 6
  AE related to other study procedure | 0
  AE leading to treatment discontinuation | 1
  AE related to TG4050 and leading to treatment discontinuation | 0
  Serious Adverse Event | 1
  Serious Adverse Event related to TG4050 | 0
  Grade 3/4 AE | 0
  Fatal AE | 1
  Fatal AE related toTG4050 | 0

2. Secondary Outcome: CA-125 Response According to GCIC
Description: Percentage of patients with a minimum 50% reduction in CA-125 serum levels lasting for 28 days relative to pre-treatment CA-125 (Carbohydrate Antigen 125) serum level per the GCIC criteria (the Gynecological Cancer Intergroup).
Time Frame: Up to 1 year. CA-125 response assessment every 3 weeks from the start of study treatment until treatment discontinuation.
Population: Safety Analysis Set (SAF): all patients who received at least one dose of TG4050
Measure: Count of Participants; unit: Participants
Arm/Group | TG4050 Arm
Number analyzed (Participants) | 6
Participants | 1

3. Secondary Outcome: Tumor Response According to RECIST 1.1
Description: Best overall response according to RECIST 1.1 was assessed for all patients, defined as follows:
  Complete Response (CR): Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Starting on Day 43 and then every nine weeks thereafter, until disease progression (estimated 12 months).
Population: Safety Analysis Set (SAF): all patients included and who received at least one dose of TG4050.
Measure: Count of Participants; unit: Participants
Arm/Group | TG4050 Arm
Number analyzed (Participants) | 6
Participants
  Stable disease | 3
  Progressive disease | 3

4. Secondary Outcome: Time to Measurable Relapse/Progression Per RECIST 1.1
Description: Time to measurable relapse/progression per RECIST 1.1 (months) is defined as the time from the date of the first treatment injection until relapse or documented progressive disease, whichever occurs first, as assessed using CT scan or MRI.
Time Frame: 43 days after treatment, and thereafter every 9 weeks until disease progression or relapse (estimated 12 months).
Population: Safety Analysis Set (SAF): all patients who received at least one dose of TG4050
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | TG4050 Arm
Number analyzed (Participants) | 6
months | 2.5 [1.4 to 11.6]

5. Secondary Outcome: Failure to Provide Rate
Description: Percentage of consented participants who could not be enrolled in the TG4050 treatment period due to manufacturing failure.
Time Frame: From informed consent (ICF) signature up to baseline.
Population: Population of participants at baseline: 37 screen failures and 6 treated.
Measure: Count of Participants; unit: Participants
Groups:
- Screened Patients: The number of patients at baseline
Arm/Group | Screened Patients
Number analyzed (Participants) | 43
Participants | 3

ADVERSE EVENTS:
Time Frame: Up to 1 year . Adverse events were collected from treatment initiation weekly for the first six weeks, every three weeks thereafter until 30 days after the last treatment administration.
Description: Adverse events (AEs) were summarized and presented by system organ class and preferred term for all participants who received at least one dose of the study treatment.
Arm/Group | TG4050 Arm
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TG4050 Arm (N=6)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) — The serious adverse event is not related to the treatment
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TG4050 Arm (N=6)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Injection site erythema (General disorders) | 5 (13)
Injection site pain (General disorders) | 3 (11)
Injection site mass (General disorders) | 2 (7)
Fatigue (General disorders) | 2 (3)
Asthenia (General disorders) | 1 (3)
Injection site irritation (General disorders) | 1 (2)
Chills (General disorders) | 1 (1)
Injection site nodule (General disorders) | 1 (1)
Injection site pruritus (General disorders) | 1 (1)
Injection site swelling (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (2)
Blood creatinine increased (Investigations) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to challenges in patient accrual, the expected sample size was not reached, rendering the originally planned secondary objectives irrelevant given the limited number of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT03839524/Prot_000.pdf
  • Statistical Analysis Plan (2025-06-10): https://cdn.clinicaltrials.gov/large-docs/24/NCT03839524/SAP_001.pdf